CLINICAL TRIAL: NCT00998322
Title: A Phase 2 Study of REOLYSIN in Combination With Gemcitabine for Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: A Study of REOLYSIN® in Combination With Gemcitabine in Patients With Advanced Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 017
Record Dates: First submitted 2009-10-15; First posted 2009-10-20 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: metastatic; pancreatic; adenocarcinoma; REOLYSIN; chemotherapy; gemcitabine
MeSH Terms: conditions — Neoplasm Metastasis; Adenocarcinoma | interventions — reolysin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN — 1E10 TCID50, 1-hour intravenous infusion on Days 1 and 2 and then Days 8 and 9 of a 21-day cycle.
Drug: Gemcitabine — 800 mg/m2 30-min infusion on Days 1 and 8 of a 21-day cycle.
  Other Names: Gemzar

SUMMARY:
The purpose of this Phase 2 study is to investigate whether intravenous administration of REOLYSIN therapeutic reovirus in combination with gemcitabine is effective and safe in the treatment of patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer remains one of the most lethal cancers, ranking as the fourth leading cause of cancer death for both men and women. The American Cancer Society estimates that 37,170 men and women (18,830 men and 18,340 women) will be diagnosed with pancreatic cancer and 33,370 men and women will die of pancreatic cancer in 2008.

Activating KRAS mutations are the most frequent genetic abnormalities in pancreatic cancer (occurring in 75% to 95% of patients).

REOLYSIN has been demonstrated to kill a wide variety of cells with mutations along the RAS pathway, including pancreatic cancer cells.

The Phase 2 study is designed to characterize the efficacy and safety of REOLYSIN given intravenously in combination with gemcitabine every 3 weeks in patients with advanced pancreatic cancer.

Response is a primary endpoint of this trial. Tumors will be evaluated by CT scan within 14 days of starting treatment, then at 6 weeks, and then every 6 weeks thereafter.

The safety of the gemcitabine and REOLYSIN combination will be assessed by the evaluation of the type, frequency and severity of adverse events, changes in clinical laboratory tests, immunogenicity and physical examination.

Patients may continue to receive therapy under this protocol, provided he/she has not experienced either progressive disease or unacceptable drug-related toxicity that does not respond to either supportive care or dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* have advanced or metastatic pancreatic adenocarcinoma who have not previously received any chemotherapy or biotherapy. Patients who have received radiotherapy with or without radiotherapy enhancers (such as low dose 5-FU) will be eligible.
* have evidence of measurable disease. However, lesions in a previous radiation field are considered non-evaluable for response. Therefore, patients must have a measurable lesion that is not in a previously irradiated field to be eligible.
* have NO continuing acute toxic effects (except alopecia) of any prior radiotherapy or surgical procedures, i.e., all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 3.0) Grade ≤1. Surgery (except biopsies) must have occurred at least 28 days prior to study enrolment.
* have received NO radiotherapy within 28 days prior to receiving study drug.
* have an ECOG Performance Score ≤ 2.
* have a life expectancy of at least 3 months.
* absolute neutrophil count (ANC) ≥ 1.5 x 10^9 [SI units 10^9/L]; Platelets ≥ 100 x10^9 [SI units 10^9/L] (without platelet transfusion); Serum creatinine ≤ 1.5 x ULN; Bilirubin ≤ 1.5 x ULN; AST/ALT ≤ 2.5 x ULN (≤ 5 x ULN if patients have liver metastasis).
* negative pregnancy test for females of childbearing potential.

Exclusion Criteria:

* no concurrent therapy with any other investigational anticancer agent while on study.
* have a history of or current evidence of brain metastasis(es).
* be on immunosuppressive therapy; have known HIV infection or active hepatitis B or C.
* be a pregnant or breast-feeding woman.
* have clinically significant cardiac disease.
* have dementia or altered mental status that would prohibit informed consent.
* have any other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Determine the clinical benefit rate (Complete Response (CR) + Partial Response (PR) + Stable Disease (SD))in the study population | 4 weeks

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the treatment regimen in the study population as measured by adverse events associated with the study treatment, and defined by established criteria. | Within 30 days of last dose of REOLYSIN
Determine the progression-free survival of this combination in patients with advanced or metastatic pancreatic adenocarcinoma. | 9-12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Montefiore Medical Center, New York, New York
  - Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas